CLINICAL TRIAL: NCT02140099
Title: Evaluation of the Healthy Relationships Plus Program for Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: CAMH Foundation (Other)
Responsible Party: Principal Investigator, David Wolfe, PhD, PhD, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 146/2013
Record Dates: First submitted 2014-05-13; First posted 2014-05-16 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Mental Health Wellness 1
Keywords: Mental health; Violence; Substance use; Adolescent; Prevention
MeSH Terms: conditions — Psychological Well-Being; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Relationships Education/Skills (Experimental): The experimental intervention is the group-based, 15-session Healthy Relationships Plus Program (HRPP). In this study, the HRPP will be offered in a condensed 8-day format (July 8-11 and 14-17, 2014). On days 1 to 7, participants will attend the program for 2 hours, and on day 8, participants will attend the program for 1 hour. The program will be facilitated by high school teachers. Eight HRPP groups will run concurrently during the study period.
  Interventions: Behavioral: Healthy Relationships Plus Program (HRPP)
- Classroom Activities (Other): The control condition is a group-based, 15-session program focusing on typical Classroom Activities. The primary activity is to create a school welcome packet for incoming Grade 9 students, with other activities including reading and physical exercise. The control condition will be offered on 8 consecutive weekdays (July 8-11 and 14-17, 2014). On days 1 to 7, participants will attend the control program for 2 hours, and on day 8, participants will attend the control program for 1 hour. The control group will be facilitated by bachelor's level research assistants and pre-service teachers. Eight control groups will run concurrently during the study period.
  Interventions: Behavioral: Control Condition (Classroom Activities)

INTERVENTIONS:
Behavioral: Healthy Relationships Plus Program (HRPP) — The Healthy Relationships Plus Program (HRPP) is an out-of-school time program that is facilitated by a teacher or other youth leader. HRPP sessions use interactive teaching strategies to discuss healthy relationships, dating violence, personal values/boundaries, communication skills, emotional health and well-being, and helping friends.
  Arms: Healthy Relationships Education/Skills
Behavioral: Control Condition (Classroom Activities)
  Arms: Classroom Activities

SUMMARY:
Adolescent risk behaviours, such as violence and substance use, are prevalent public health concerns in Canada. Further, these behaviours often co-occur, and are associated with poor mental health. However, the majority of prevention programs focus on preventing single issues and do not consider mental health, and also neglect the importance of relationships when promoting positive youth development. To address this gap, the Centre for Addiction and Mental Health (CAMH) Centre for Prevention Science designed the Fourth R Healthy Relationships Plus Program, a small group program focused on the promotion of positive mental health and the reduction of violence and substance use, via the development of improved communication, interpersonal and help-seeking skills. The purpose of this study is to evaluate the Fourth R Healthy Relationships Plus program using both outcome (randomized controlled trial design with follow-up at pre-test, post-test, and 4, 8 and 12 months) and process evaluation tools.

The primary study hypothesis is that participation in the Fourth R Healthy Relationships Plus program will be associated with positive growth in treatment participants' psychological well-being from pre-test to 12-month follow-up, as compared to control participants. In secondary analyses, the study will explore if treatment participants report less substance use, peer violence, bullying and dating violence at 12-month follow-up than control participants. Since certain person-level (e.g., sex, personality, executive functioning) and program-level (e.g., implementation quality) variables may moderate treatment-outcome relationships, these associations will also be explored. The final hypothesis is that treatment participants will report better attitudes, knowledge and assertive communication at post-test compared to control participants, and that these improvements will mediate the association between program participation and 12-month outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled (as of March 2014) in grade 9 or 10 at schools serving as study sites

Exclusion Criteria:

* Not available during the period July 7-17, 2014 (the main study period)
* Not interested in participating in the project, as assessed on study information form
* Identified by the Guidance Office at his/her school as posing a serious safety risk to him/herself or others

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 238 (Actual)
Dates: Start 2014-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Growth from baseline to 12-month follow-up on a multi-variable latent psychological well-being construct | Baseline, Month 4, Month 8, Month 12
  Scales included to indicate the latent psychological well-being construct are:
  1. hope
  2. purpose
  3. depression/anxiety
  4. emotion regulation
  5. coping behaviours
  6. flourishing mental health

SECONDARY OUTCOMES:
Decrease in reported perpetration on the Conflict in Adolescent Dating Relationships Inventory (CADRI) Physical Abuse and Threatening Behaviour sub-scales in treatment versus control participants at 12 month follow-up, compared to baseline | Baseline, Month 12
Decrease in reported perpetration on the Cyber Dating Abuse scale in treatment versus control participants at 12 month follow-up, compared to baseline | Baseline, Month 12
Decrease in reported physical fighting in treatment versus control participants at 12 month follow-up, compared to baseline | Baseline, Month 12
Decrease in past 30 day drinking frequency in treatment versus control participants at 12 month follow-up, compared to baseline | Baseline, Month 12
Decrease in past 30 day heavy episodic drinking (binge drinking) in treatment versus control participants at 12 month follow-up, compared to baseline | Baseline, Month 12
Decrease in past 30 day marijuana use in treatment versus control participants at 12 month follow-up, compared to baseline | Baseline, Month 12
Decrease in reported likelihood to try illicit drugs (e.g., marijuana; other illegal drugs; non-prescribed prescription drugs) during the next 12 months in treatment versus control participants at 12 month follow-up, compared to baseline | Baseline, Month 12
Decrease in reported perpetration on the Bullying Evaluation and Strategies Tool (grade 7-12 items) in treatment versus control participants at 12 month follow-up, compared to baseline | Baseline, Month 12
Decrease in hostility on a 4-point hostility scale in treatment versus control participants at 10 days, compared to baseline | Baseline, Day 10
Improvement in drug attitudes on the 4-point Drug Attitude Scale in treatment versus control participants at 10 days, compared to baseline | Baseline, Day 10
Improvement in attitudes towards violence on the 4-point Acceptability of Violence scale in treatment versus control participants at 10 days, compared to baseline | Baseline, Day 10
Greater use of program concepts in written responses to 3 open-ended knowledge questions in treatment versus control participants at 10 days. | Day 10
Improvement in interpersonal negotiation strategy scores with parents in treatment versus control participants at 10 days, compared to baseline | Baseline, Day 10
Improvement in interpersonal negotiation strategy scores with peers in treatment versus control participants at 10 days, compared to baseline | Baseline, Day 10
Improvement in interpersonal negotiation strategy scores with romantic partners in treatment versus control participants at 10 days, compared to baseline | Baseline, Day 10

OTHER OUTCOMES:
Growth from baseline to 12-month follow-up on psychological well-being in male vs. female participants | Baseline, Month 4, Month 8, Month 12
  We plan subgroup analyses by sex to investigate if males' and females' psychological well-being differs over follow-up period. We have no a priori assumptions about sex differences.

CONTACTS AND LOCATIONS:
Overall Officials: David A Wolfe, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- CAMH Centre for Prevention Science, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiodo D, Crooks CV, Wolfe DA, McIsaac C, Hughes R, Jaffe PG. Longitudinal prediction and concurrent functioning of adolescent girls demonstrating various profiles of dating violence and victimization. Prev Sci. 2012 Aug;13(4):350-9. doi: 10.1007/s11121-011-0236-3. PMID 21769657
- [Background] Wolfe DA, Crooks CV, Chiodo D, Hughes R, Ellis W. Observations of adolescent peer resistance skills following a classroom-based healthy relationship program: a post-intervention comparison. Prev Sci. 2012 Apr;13(2):196-205. doi: 10.1007/s11121-011-0256-z. PMID 22057307
- [Background] Crooks CV, Scott K, Ellis W, Wolfe DA. Impact of a universal school-based violence prevention program on violent delinquency: distinctive benefits for youth with maltreatment histories. Child Abuse Negl. 2011 Jun;35(6):393-400. doi: 10.1016/j.chiabu.2011.03.002. Epub 2011 Jun 8. PMID 21652072
- [Background] Wolfe DA, Crooks C, Jaffe P, Chiodo D, Hughes R, Ellis W, Stitt L, Donner A. A school-based program to prevent adolescent dating violence: a cluster randomized trial. Arch Pediatr Adolesc Med. 2009 Aug;163(8):692-9. doi: 10.1001/archpediatrics.2009.69. PMID 19652099
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto. — http://www.camh.ca/en/research
- See also: CAMH Centre for Prevention Science and Fourth R homepage — http://www.youthrelationships.org